CLINICAL TRIAL: NCT03513237
Title: Routine Cervical Dilatation at the Non-labor Caesarean Section and Its Influence on Postoperative Pain: A Randomised Controlled Trial
Brief Title: Routine Cervical Dilatation at the Non-labour Caesarean Section and Its Influence on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Routine cervical dilatation
Record Dates: First submitted 2018-03-24; First posted 2018-05-01 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Labor Stage, First

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The women will be blinded to the intervention, but the investigator will not be blinded to the procedure allocation (due to the nature of the intervention).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical dilation group (Experimental): the surgeon will perform the cervical dilatation by inserting the double-gloved index ﬁnger into the cervical canal after extraction of placenta and membranes and will remove the outer gloves after digital dilatation of the cervix.
  Interventions: Procedure: Cervical dilation
- no cervical dilation group (No Intervention): No cervical dilation will be done.

INTERVENTIONS:
Procedure: Cervical dilation — manual dilatation of the cervix using surgeon's finger.
  Arms: Cervical dilation group

SUMMARY:
Caesarean section is a common method of delivery in obstetrics. With the recent increase in the rate of this procedure, it is wise to understand and implement the optimal surgical technique. Therefore, different operational methods have been defined to reduce the risk of peri/post-operative morbidity.

The digital dilatation of cervix during elective caesarean section has still been a concern when evaluating this issue. This procedure is supposed to help the drainage of blood and lochia postpartum, thus reducing infection or the risk of postpartum haemorrhage (PPH). However, on the contrary, this mechanical manipulation may also result in contamination by a vaginal micro-organism and increase the risk of infections or cervical trauma. Additionally, the effect of routine cervical dilatation on patients' perception of pain has not been studied sufficiently yet. As a result, the current literature lacks evidence of cervical dilatation on postoperative pain and is even not all in agreement regarding the potential benefits on overall maternal morbidity.

DETAILED DESCRIPTION:
Caesarean section is a common method of delivery in obstetrics. With the recent increase in the rate of this procedure, it is wise to understand and implement the optimal surgical technique. Therefore, different operational methods have been defined to reduce the risk of peri/post-operative morbidity.

The digital dilatation of cervix during elective caesarean section has still been a concern when evaluating this issue. This procedure is supposed to help the drainage of blood and lochia postpartum, thus reducing infection or the risk of postpartum haemorrhage (PPH). However, on the contrary, this mechanical manipulation may also result in contamination by a vaginal micro-organism and increase the risk of infections or cervical trauma. Additionally, the effect of routine cervical dilatation on patients' perception of pain has not been studied sufficiently yet. As a result, the current literature lacks evidence of cervical dilatation on postoperative pain and is even not all in agreement regarding the potential benefits on overall maternal morbidity.

In this prospective study, our primary aim is to evaluate the effect of intra-operative digital dilatation of cervix on post-operative pain. We hypothesize that dilatation of the cervix as compared with non-dilatation will result in less pain by reducing fluid and blood stasis inside the uterine cavity. Our secondary objective is to assess the maternal morbidity including a reduction in haemoglobin concentrations, puerperal fever, puerperal endometritis and wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Gestational age: ≥ 37 weeks gestation with a BMI > 25 kg/m².
* Singleton pregnancy.
* Free medical history.
* Nulliparous women who would undergo their ﬁrst elective cesarean section at term without any labor pain or multiparous women who had undergone cesarean section in all the previous pregnancies without any labor pain.)

Exclusion Criteria:

* the onset of labor with dilation of the cervix or women who felt labor pain before their previous cesarean operations.
* Prolonged premature rupture of membranes.
* Fever on admission or ongoing infection as Chorioamnionitis.
* Current antibiotic therapy.
* The need for Blood transfusion during or after CS.
* Emergency CS and preterm cesarean section.
* Pre-existing maternal disease as prepregnancy diabetes mellitus.
* Women at term who had risk factors for postpartum haemorrhage, e.g. placenta previa
* Women with Chronic pelvic pain

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
mean change of postoperative pain over time points mentioned in the time frame | 8th, 24th, and 48th hours ,4th and 7th day after the operation
  will be assessed using Numerical Rating Scale which is a segmented numeric version of the visual analog scale (VAS) in which the patient selects a whole number (0-10 integers) that best reflects the intensity of her pain.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").the numeric rating scale will be either administered verbally (therefore also by telephone) or graphically for self-completion.Scores range from 0-10 points, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Puerperal Endometritis | 48 hours after operation
  body temperature higher than 38.5 Celsius degree with concomitant foul-smelling discharge or abnormally tender uterus on bimanual examination
puerperal fever | 1st and 2nd day postoperative
  a persistent fever of at least 38 Celsius degree taken from the axillary region on two occasions more than 6 h apart after the ﬁrst postpartum day and not associated with lower abdominal or pelvic tenderness and no signs of infection elsewhere.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Ahmed Samy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alalfy M, Yehia A, Samy A. Routine cervical dilatation at caesarean section and its influence on postoperative pain and complications in obese women: a double blind randomized controlled trial. J Matern Fetal Neonatal Med. 2021 Jun;34(12):1906-1913. doi: 10.1080/14767058.2019.1651274. Epub 2019 Aug 11. PMID 31401929